CLINICAL TRIAL: NCT02264457
Title: A Randomised Intra-patient Comparison of Closed Loop and Plate Haptic Toric, Aspheric, Aberration Neutral, Hydrophilic Acrylic Intraocular Lenses in Patients With Bilateral Astigmatism
Brief Title: A Intra-patient Comparison of Closed Loop and Plate Haptic Toric Intraocular Lenses
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Plymouth (Other)
Collaborators: BMI Southend Hospital (Other)
Responsible Party: Principal Investigator, Dr Phillip J Buckhurst, Associate Professor (Senior Lecturer), University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IISR-2014-003
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Cataract
Keywords: Lenses, Intraocular
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- First eye closed loop haptic (Other): subjects implanted with the Closed loop haptic during first eye surgery and the plate haptics toric intraocular lens during second eye surgery
  Interventions: Device: T-flex Aspheric Toric IOL; Device: AT TORBI toric IOL
- First eye plate haptic (Other): subjects implanted with the plate haptic toric during first eye surgery and the closed loop haptic toric intraocular lens during second eye surgery
  Interventions: Device: T-flex Aspheric Toric IOL; Device: AT TORBI toric IOL

INTERVENTIONS:
Device: T-flex Aspheric Toric IOL
Device: AT TORBI toric IOL

SUMMARY:
During cataract surgery an artificial lens is implanted in the eye. These artificial lenses are called intraocular lenses (IOLs) and there are many different types of IOL designs. Your eyes have astigmatism, which is a normal and common characteristic of the eye. If left uncorrected the astigmatism would mean that you would need to wear spectacles for viewing distance objects. New IOL designs called toric IOLs help to correct the astigmatism to improve your vision after cataract surgery. This study has been designed to look at how well a toric IOL corrects this astigmatism so that you do not need to wear spectacles for viewing distance objects. There are many designs of these toric IOLs and for this study we are looking to compare two different designs of toric IOLs by putting one lens in your right eye and a different type of lens in your left eye. Both lenses are commercially available and are commonly implanted IOLs. Using new non-invasive methods we hope to be able to better judge the visual performance of these lenses and the ability of these lenses to correct astigmatism. In addition the study will involve imaging and examining the IOLs to determine the prevalence of any post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years, bilateral significant corneal astigmatism >1.50D.
* Requiring a Toric IOL within the following power range:
* Sphere +6.00D to +30.00D
* Cylinder +1.00D to +6.00D

Exclusion Criteria:

* Amblyopia,
* predicted bilateral post-op corneal astigmatism of <1.50D,
* irregular astigmatism,
* dilated pupil size smaller than 5mm,
* macular pathology,
* glaucoma,
* retinal disease,
* corneal disease,
* abnormal iris,
* pupil deformation and
* any previous corneal or intraocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity | Visit 1 (1-2 days post implantation), visit 2 (1-2 weeks post implantation), visit 3 (1-2 months post implantation) and visit 4 (3-4 months

SECONDARY OUTCOMES:
Manifest refraction | Visit 1 (1-2 days post implantation), visit 2 (1-2 weeks post implantation), visit 3 (1-2 months post implantation) and visit 4 (3-4 months)
Rotational stability | Visit 1 (1-2 days post implantation), visit 2 (1-2 weeks post implantation), visit 3 (1-2 months post implantation) and visit 4 (3-4 months)
IOL centration | Visit 1 (1-2 days post implantation), visit 2 (1-2 weeks post implantation), visit 3 (1-2 months post implantation) and visit 4 (3-4 months)
Prevalence of posterior capsular Opacification | visit 4 (3-4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip J Buckhurst, PhD, Principal Investigator — Plymouth University
Locations (1):
- BMI Southend Private Hospital, Westcliff-on-Sea, Essex, United Kingdom